CLINICAL TRIAL: NCT04265014
Title: Comparison of Goal-directed and Liberal Fluid Management With Minimal Invasive Hemodynamic Monitoring in Abdominal Surgeries: A Randomized Prospective Study
Brief Title: Comparison of Goal-directed and Liberal Fluid Management
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: we didn't have any patient
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 165/2017
Record Dates: First submitted 2020-01-28; First posted 2020-02-11 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Goal-Directed Fluid Therapy; Hemodynamic Monitoring; Fluid Management

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Goal-directed fluid treatment (Active Comparator): Fluid management will be performed according to SVV and CI monitoring. When patients have SVV>10%, 250 cc crystalloid will be administered and when SVV fell below 10% during 30-minute monitoring standard (5 mL/kg/hr) crystalloid infusion continues. If SVV continues above 10%, a second fluid bolus of 250 cc colloid (minifluid challenge) will be administered.
  If the desired SVV level can not be reached, the Hct values will be examined. Blood replacement will be performed when Hct<30% in patients with coronary artery disease (CAD) and when Hct<25% for other patient groups. If the desired SVV level can not be reached in spite of blood replacement products, if CI will be below 2.5 L/min/m2 vasopressor will begun. If SVV will be at normal values with CI below 2.5 L/min/m2, inotrop will begun.
  Interventions: Other: Goal-directed fluid treatment
- liberal fluid treatment (Active Comparator): Fluid management will be performed according to MAP, HR and urine output.
  If peroperative urine amounts will be <0.5 mL/kg/hr during two-hour monitoring, with MAP<65 mmHg, HR>100/min for at least 30 minutes and CVP falls 20% compared to basal values, the same anesthesiologist will begin additional fluid replacement of 5 mL/kg/hr based on clinical experience.
  Blood product replacement will be provided at Hct<30% for those with coronary artery disease and at Hct<25% for other patients.
  Interventions: Other: Liberal Fluid Therapy

INTERVENTIONS:
Other: Goal-directed fluid treatment — Goal-directed fluid treatment for major abdominal surgery
  Arms: Goal-directed fluid treatment
Other: Liberal Fluid Therapy — Liberal Fluid Therapy for major abdominal surgery
  Arms: liberal fluid treatment

SUMMARY:
Background: The investigators aim is to indicate that the "goal directed fluid management" is more effective for open abdominal surgeries by performing perioperative hemodynamic monitorisation using a minimal invasive pulse counter analysis method.

Methods: The study will be included 90 participants with ASA II-III risk score aged from 18-64 years. The prospective and randomized participants will be divided into 2 groups as liberal (Group L) and goal-directed fluid therapy (Group G) fluid treatment. Hemodynamic parameters and arterial blood gas analysis will be recorded at 30 min intervals. Preoperative and postoperative creatinine values, CR-POSSUM physiological score, Charlson comorbidity index (CCI), perioperative and postoperative vasopressor use, postoperative acute kidney injury network (AKIN), postoperative intensive care requirements, duration of hospital stay and 30-day mortality will be recorded.

DETAILED DESCRIPTION:
Blood will be taken and assessed from the participants preoperatively one day before surgery and creatinine, neutrophil, lymphocyte and neutrophil / lymphocyte values will be recorded.

Though the gastrointestinal surgery team is the same, randomization will not be applied for the primary operating surgeon and primary surgeon selection will not be performed. Participants in both groups will have age, gender, height, weight, body mass index (BMI), comorbidities, CCI, POSSUM physiologic score and ASA risk score recorded. After being taken to the operation room, standard monitoring (ECG, SO2, NIBP) will be performed. A peripheral venous route will be opened with an 18-gauge needle. Participants will be began 5 mL/kg/hr crystalloid (isolyte) infusion as standard. Later participants who accept will have an epidural catheter inserted at the thoracic 10-11 level. After ensuring hemodynamic stabilization in both groups, sedation will be provided with 0.03 mg/kg midazolam and arterial monitoring will be provided with radial artery cannulation with a 20-gauge peripheral cannula.

Induction and General Anesthesia Management:

For induction 1-2 mcg/kg fentanyl, 2 mg/kg propofol and 0.6 mg/kg rocuronium will be used, and participants will be orotracheally intubated after two minute ventilation. A MAQUET flow-I anesthesia device will be placed in volume control (VC) mode by setting to 8 mL/kg tidal volume and 12/min respiratory count according to ideal body weight with PetCO2 35-45 mmHg. Later, central venous catheterization will be performed on the right internal jugular vein using USG guidance. Sevoflurane (MAC 0.7-0.9) and remifentanil infusion (0.05-0.3 mcg/kg/min) will be used in anesthesia maintenance.

Monitoring:

After radial artery and central jugular vein catheterization in Group G, they will be linked to an EV1000 Flo-trac monitor and monitoring provided continuous mean arterial pressure (MAP) monitoring with heart rate (HR), stroke volume variation (SVV), central venous pressure (CVP), systemic vascular resistance index (SVRI) and cardiac index (CI) measured every minute. After monitoring blood gas will be taken and the initial value accepted as time-1 (t1). At 5 minute intervals, mean arterial pressure (MAP), momentary heart rate (HR) will be recorded, with CVP, CI, SVV, and SVRI recorded at 30 minute intervals for a total of 240 minutes (t1, t2, t3, t4, t5, t6, t7, t8, t9), urine amount and blood gas values (pH, PCO2, PO2, bicarbonate (HCO3), base minus (BM), lactate (lac), hemoglobin (Hb), hematocrit (Ht)) will also be recorded.

In Group L, radial arterial cannulation and central jugular venous catheterization will be performed with the first value during monitoring accepted as t1. Then HR and MPA will be recorded at 5-minute intervals, CVP at 30 minute intervals for a total of 240 minutes (t1, t2, t3, t4, t5, t6, t7, t8, t9) and urine amount and blood gas values (pH, PCO2, PO2, HCO3, BM, lac, Hb, Ht) will also be recorded.

Peroperative fluid management:

1. Group G:

   Fluid management will be performed according to SVV and CI monitoring. When participants have SVV>10%, 250 cc crystalloid will be administered and when SVV fell below 10% during 30-minute monitoring standard (5 mL/kg/hr) crystalloid infusion continues. If SVV continues above 10%, a second fluid bolus of 250 cc colloid (minifluid challenge) will be administered. If the desired SVV level can not be reached, the Hct values will be examined. Blood replacement will be performed when Hct<30% in participants with coronary artery disease (CAD) and when Hct<25% for other groups. If the desired SVV level can not be reached in spite of blood replacement products, if CI will be below 2.5 L/min/m2 vasopressor will begun. If SVV will be at normal values with CI below 2.5 L/min/m2, inotrop will begun.
2. Group L:

Fluid management will be performed according to MAP, HR and urine output. If peroperative urine amounts will be <0.5 mL/kg/hr during two-hour monitoring, with MAP<65 mmHg, HR>100/min for at least 30 minutes and CVP falls 20% compared to basal values, the same anesthesiologist will begin additional fluid replacement of 5 mL/kg/hr based on clinical experience. Blood product replacement will be provided at Hct<30% for those with coronary artery disease and at Hct<25% for other participants.

The operation durations, administered fluid types, fluid amounts and blood product amounts will be recorded. Participants having intensive care need preoperatively planned intensive care will have planned admission, while participants developing hemodynamic instability linked to peroperative surgery or anesthesia will be admitted as unplanned care. All participants will have creatinine, neutrophil, lymphocyte and neutrophil/lymphocyte values recorded in the 1st and 24th hours postoperative and participants with fever (>38 °C) in the 1st day will be recorded. Acute kidney injury network (AKIN) classification will be made according to creatinine values measured preoperatively and on the postoperative 1st day. In the postoperative 30-day period, duration of hospital stay, surgical and pulmonary complications, inotrop or vasopressor requirements, reason for admission to intensive care, and duration of stay in intensive care if required will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients with major abdominal surgery
* ASA risk classification II-III

Exclusion Criteria:

* Peripheral artery disease
* Not in sinus rhythm
* Peroperative major hemorrhage (more than 500 mL hemorrhage within 1 hour)
* Pregnant or breastfeeding
* Advanced degree of liver and renal failure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Peroperative Hemodiynamic, Mean Arterial Pressure | During the surgery
  Mean arterial pressure (mmHg)
Peroperative Hemodiynamic, Kidney Function | During the surgery
  Urine output (ml/h)
Peroperative Hemodiynamic, Pulse | During the surgery
  Heart rate (beats per minute)
Peroperative Hemodiynamic, Fluid response | During the surgery
  Stroke Volume Variation (%)
Peroperative Hemodiynamic, Cardiac output | During the surgery
  Cardiac Index (l/min/m2)

SECONDARY OUTCOMES:
Number of Participants | 5 months
  The study will be terminated when a total of 90 patients are reached.

CONTACTS AND LOCATIONS:
Locations (1):
- Bakırkoy Sadi Konuk Training and Research Hospital, Istanbul, Turkey (Türkiye)